CLINICAL TRIAL: NCT04600219
Title: The Effect of Tyrosine Kinase Receptor Axl on Dialysis Prognosis in Chronic Hemodialysis Patients: a Cohort Study
Brief Title: The Effect of Tyrosine Kinase Receptor Axl on Dialysis Prognosis in Chronic Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the department of Nephrology,Shanghai 10th people's hospital, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: AHD2020
Record Dates: First submitted 2020-10-21; First posted 2020-10-23 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hemodialysis Complication
Keywords: hemodialysis; Axl; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate whether tyrosine kinase receptor Axl affects the dialysis prognosis in chronic hemodialysis patients

DETAILED DESCRIPTION:
It is reported that hemodialysis (HD) patients often develop chronic systemic inflammatoion, and increased inflammatory activity is associated with vascular access failure, cardiovascular disease and death in HD patients. The interaction of Axl and its ligand Gas6 plays an important role in modulating immune response, inhabiting toll-like receptor (TLR) signaling and suppressing inflammatory cytokines production. Thus, we want to investigate the relationship between tyrosine kinase receptor Axl and the dialysis prognosis in HD patients in three-years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis for more than 6 months

Exclusion Criteria:

* patients who received warfarin therapy;
* patients with chronic infectious disease or acute infection;
* patients with hemodialysis inadequacy;
* the age of patients is older than 65 years or younger than 18 years.
* patients who can not sign an informed consent or disagree to follow up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients undergoing hemodialysis treatment
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
death | 3 years
  death
dialysis complication | 3 years
  vascular access failure, stroke, acute coronary syndrome, heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, MD,PhD, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No